CLINICAL TRIAL: NCT04443790
Title: Obesity Control Through Leptogenic Drugs
Brief Title: Clinical Evaluation of Polyherbal Coded Formulation Obesecure for Leptin Regulation and Obesity Management
Acronym: CEOLO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hafiz Muhammad Asif (Other)
Collaborators: Hamdard University (Other); Government College University Faisalabad (Other)
Responsible Party: Sponsor-Investigator, Hafiz Muhammad Asif, Clinical Trials Registrar for Shifaulmulk, Shifa Ul Mulk Memorial Hospital
Organization: Shifa Ul Mulk Memorial Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCUF/ERC/1817
Record Dates: First submitted 2020-06-19; First posted 2020-06-23 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Leptin Deficiency; Obesity
MeSH Terms: conditions — Obesity, Morbid; Obesity

STUDY DESIGN:
Intervention Model Description: Multicentre, two arm parallel randomized controlled clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Obesecure Capsules (Test Group) (Active Comparator): A dose of 500mg capsule twice daily of Polyherbal formulation Obesecure was given in the test group for three months. Short term effectiveness was assessed by BMI calculation on follow up visit after two weeks and long term follow up was assessed by BMI and Leptin Level at three months.
  Interventions: Drug: Leptin Human
- Plasicure (Control Group) (Placebo Comparator): A dose of 500mg capsule twice daily of Placebo as Plasicure was given in the control group for three months. Short term effectiveness was assessed by BMI calculation on follow up visit after two weeks and long term follow up was assessed by BMI and Leptin Level at three months.
  Interventions: Drug: Leptin Human

INTERVENTIONS:
Drug: Leptin Human
  Other Names: Obesecure

SUMMARY:
The study was designed to explore an alternative approach to reduce weight in human beings using a polyherbal formulation. A polyherbal formulation named as Obesecure was developed after screening of local medicinal flora. The formulation was further improved after pilot studies and Phase-I Clinical Trials.

DETAILED DESCRIPTION:
Obesity is a common disease of developing countries including Pakistan. Obesity is a risk factor for many diseases which can be life-threatening or making the person unable to perform daily routine work. Obesity is considered a risk factor for different diseases like cardiovascular diseases, hormonal imbalance, infections, malignancies and chest problems. The leptin hormone has appetite suppressing and energy dissipation activity in the body. A screening study on animals was carried out to find out the leptin enhancing medicinal plants from locally available plants in Pakistan. This study was aimed to see the combined effects of the Leptogenic drug Obesecure on weight management.

Patients of age20 to 50 years with BMI more than 25, not taking any anti-obesity drugs one-month prior to start of study were enrolled. The Participants were randomly allocated to receive either Obesecure or placebo twice a day for three months in Shifa-ul-mulk Hospital, PRIEM Health Care Clinic (Pakistan) and Ria Eastern Medicine Clinic (Pakistan).

An acute toxicity study showed no adverse effect of taking Obesecure prior to clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of age20 to 50 years with BMI more than 25
2. Only those participants were included who were willing
3. Patients of any marital status were included
4. Only those participants were included who did not take any antiobesity drug one-month prior to start of study

Exclusion Criteria:

1. Taking an anti-obesity drug in the previous month
2. Pregnant
3. Allergic to laxative drugs
4. Recurrent weight gain history after antiobesity treatment
5. Liver disease
6. Taking hormonal therapy, menopausal women
7. Diabetes mellitus
8. Cardiac problem and hypertension

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 132 (Actual)
Dates: Start 2015-04-10 (Actual); Primary Completion 2018-03-20 (Actual); Study Completion 2018-05-20 (Actual)

PRIMARY OUTCOMES:
Leptin Level | 3 months
  Appetite suppression and energy dissipation
BMI (kg/m²) at baseline | 3 Months
  weight reduction effects

CONTACTS AND LOCATIONS:
Overall Officials: Ejaz Mohiuddin, Ph.D, Study Director — Hamdard University
Locations (1):
- clinical trial was conducted in Karachi,Islamabad and Faisalabad, Karachi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
IPD will be shared to other researchers on request

REFERENCES:
- [Background] Wasim M, Awan FR, Najam SS, Khan AR, Khan HN. Role of Leptin Deficiency, Inefficiency, and Leptin Receptors in Obesity. Biochem Genet. 2016 Oct;54(5):565-72. doi: 10.1007/s10528-016-9751-z. Epub 2016 Jun 16. PMID 27313173
- [Background] Farr OM, Gavrieli A, Mantzoros CS. Leptin applications in 2015: what have we learned about leptin and obesity? Curr Opin Endocrinol Diabetes Obes. 2015 Oct;22(5):353-9. doi: 10.1097/MED.0000000000000184. PMID 26313897
- [Result] Lee JH, Lee JJ, Cho WK, Yim NH, Kim HK, Yun B, Ma JY. KBH-1, an herbal composition, improves hepatic steatosis and leptin resistance in high-fat diet-induced obese rats. BMC Complement Altern Med. 2016 Sep 13;16(1):355. doi: 10.1186/s12906-016-1265-z. PMID 27618865